CLINICAL TRIAL: NCT04971954
Title: Using Nicotine to Reverse Age-related Auditory Processing Deficits: Human Psychophysics and Electrophysiology
Brief Title: Using Nicotine to Reverse Age-related Auditory Processing Deficits
Acronym: Nicotine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Fan-Gang Zeng, Professor, University of California, Irvine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 20139964; 1R01AG067073 (NIH)
Record Dates: First submitted 2021-06-16; First posted 2021-07-22 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Auditory Perceptual Impairment; Aging
Keywords: nicotine; biomarker
MeSH Terms: conditions — Auditory perceptual impairment | interventions — Nicotine Chewing Gum

STUDY DESIGN:
Intervention Model Description: The nicotine and placebo gums will be administered in randomized, double-blind, counterbalanced fashion.
Who Masked: Participant, Investigator
Masking Description: Nicotine (6 mg) will be administered in the form of polacrilex gum that is available as an over-the-counter medication. The placebo will also be a commercially available gum that resembles the nicotine gum in flavor, size, shape, color, and texture.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nicotine gum (Experimental): Nicotine (6 mg) will be administered in the form of polacrilex gum that is available as an over-the-counter medication
  Interventions: Other: Nicotine gum
- Placebo gum (Placebo Comparator): The placebo will also be a commercially available gum that resembles the nicotine gum in flavor, size, shape, color, and texture.
  Interventions: Other: Placebo gum

INTERVENTIONS:
Other: Nicotine gum — Nicotine (6 mg) will be administered in the form of polacrilex gum that is available as an over-the-counter medication
  Arms: Nicotine gum
Other: Placebo gum — The placebo will also be a commercially available gum that resembles the nicotine gum in flavor, size, shape, color, and texture.
  Arms: Placebo gum

SUMMARY:
The present study will evaluate the effects of both aging and nicotine on psychophysical tasks and electrophysiological measures. Nicotine will be administered to study participants in the form of gum that is available as an over-the-counter medication. The hypothesis is that nicotine will reverse the detrimental effects of aging on auditory processing. The proposed experiments will characterize the effects of nicotine and may eventually lead to improved treatments of hearing loss in a variety of patient populations and in healthy aging.

DETAILED DESCRIPTION:
Study participants will be recruited in two age groups: young (18-28 years) and old (60-85). Each participant will participate in two psychophysical and electrophysiological test sessions. For each of the two sessions, the participant will be administered gum before the test. For one of these sessions, the gum will be polacrilex that contains 6-mg nicotine, and for the other session, the gum will be a placebo control. The study will be double-blind, meaning that neither the experimenter nor the participant will know whether the participant has received nicotine or placebo for a given session. The study has a cross-over design, meaning that all participants will receive both nicotine and placebo in separate sessions. Finally, the order of drug administration will be counterbalanced, meaning that equal numbers of participants will receive 1) nicotine in session one and placebo in session two, and 2) placebo in session one and nicotine in session two.

ELIGIBILITY:
Inclusion Criteria:

* between 18 and 85 years of age
* non-smokers with a score of 0-2 out of 10 maximum on the Fagerström index of smoking dependency
* cognitive performance within two standard deviations of the CERAD mean

Exclusion Criteria:

* less than 18 or greater than 85 years of age
* deafness or excessive hearing loss
* smokers with a score between 3 and 10 on the Fagerström index of smoking dependency
* history of psychiatric illness, neurological disorders, diabetes mellitus, renal failure, or cardiovascular disease
* regular use of prescription medications (excluding oral contraceptives)
* drug dependency

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Hearing thresholds | 1 hour
  Hearing thresholds in dB SPL will be measured as a function of sound frequency from 125 Hz to 8000 Hz in quiet or in noise.
Modulation detection | 1 hour
  Amplitude-modulated sounds will be presented at 70 dB SPL or a comfortable level. The detection threshold in percent modulation depth (m= 0 to 100) will be recorded and converted into signal-to-noise ratios in dB (=20log(m)).
Envelope following responses | 2 hours
  Electrophysiological responses will be recorded in response to amplitude or frequency-modulated sounds. The sounds will be presented at 70 dB SPL or a comfortable level. The EEG signal strength that is in synchrony with the modulation frequency in micro-Volts will be recorded.

SECONDARY OUTCOMES:
Heart rate | 10 minutes
  Pulse rate in pulses per minute will be measured via pulse oximetry.
Mood change | 10 minutes
  Mood change will be measured by a 9-category rating scale including: energy, contentedness, focus, relaxation, calmness, alertness, hunger etc.
Nicotine side effects | 10 minutes
  Side effects will be rated on a 5-point scale including: 1 = none (no symptoms at all); 2 = mild (slight jitters); 3 = moderate (jittery, slight dull headache); 4 = moderately severe (jittery, dull headache, mild nausea); 5 = severe (jittery, dull or pounding headache, nausea, vomiting).

OTHER OUTCOMES:
Cognition | 1 hour
  Word learning, recall and animal fluency tests from the Consortium to Establish a Registry for Alzheimer's Disease (CERAD) will be measured and normalized to the national standard distribution, with a score of 0 equaling to the mean and 1 being one standard deviation above the mean performance.

CONTACTS AND LOCATIONS:
Overall Officials: Fan-Gang Zeng, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- Hearing and Speech Lab, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pham CQ, Kapolowicz MR, Metherate R, Zeng FG. Nicotine enhances auditory processing in healthy and normal-hearing young adult nonsmokers. Psychopharmacology (Berl). 2020 Mar;237(3):833-840. doi: 10.1007/s00213-019-05421-x. Epub 2019 Dec 12. PMID 31832719
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Morris JC, Heyman A, Mohs RC, Hughes JP, van Belle G, Fillenbaum G, Mellits ED, Clark C. The Consortium to Establish a Registry for Alzheimer's Disease (CERAD). Part I. Clinical and neuropsychological assessment of Alzheimer's disease. Neurology. 1989 Sep;39(9):1159-65. doi: 10.1212/wnl.39.9.1159. PMID 2771064